CLINICAL TRIAL: NCT02728947
Title: A Single Group and Open-label Study to Evaluate Pharmacokinetic Profile of Neupro Patch Administrated at 2 mg, 4 mg, 6 mg and 8 mg/Day Weekly in Patients With Early-stage Parkinson's Disease
Brief Title: Pharmacokinetic Profile of Neupro Patch Administrated at 2 mg, 4 mg, 6 mg and 8 mg/Day Weekly in Patients With Early-stage Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LY03003-CT-USA-103
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 2mg (Active Comparator): 1 week on 2mg/24 hr patch
  Interventions: Drug: ROTIGOTINE
- 4mg (Active Comparator): 1 week on 4mg/24hr patch
  Interventions: Drug: ROTIGOTINE
- 6mg (Active Comparator): 1 week on 6mg/24hr patch
  Interventions: Drug: ROTIGOTINE
- 8mg (Active Comparator): 1 week on 8mg/24hr patch
  Interventions: Drug: ROTIGOTINE

INTERVENTIONS:
Drug: ROTIGOTINE — 1 week at each dose
  Other Names: Neupro

SUMMARY:
To study the profile of Neupro patch administrated at 2 mg, 4 mg, 6 mg and 8 mg/day weekly in patients with early-stage Parkinson's disease

DETAILED DESCRIPTION:
A single group and open-label study to evaluate pharmacokinetic profile of Neupro patch administrated at 2 mg, 4 mg, 6 mg and 8 mg/day weekly in patients with early-stage Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

1. Patient who is capable of giving informed consent and complying with study procedures
2. Patient who has Idiopathic Parkinson's Disease defined by the cardinal sign, bradykinesia, plus the presence of at least 1 of the following: resting tremor, rigidity, or impairment of postural reflexes, and without any other known or suspected cause of Parkinsonism
3. Patient who is Hoehn & Yahr stage less than or equal to 3
4. Patient who is male or female aged greater than or equal to 18 years at Screening
5. Patient who has a Mini Mental State Examination (MMSE) score of greater than or equal to 25
6. Patient who has a Unified Parkinson's Disease Rating Scale (UPDRS) motor score (Part III) of greater than or equal to 10 but less then or equal to 30 at Screening

Exclusion Criteria:

1. Patient who has atypical Parkinson's syndrome(s) due to drugs (e.g., metoclopramide, flunarizine), metabolic neurogenetic disorders (e.g., Wilson's Disease), encephalitis, cerebrovascular disease, or degenerative disease (e.g., progressive Supranuclear Palsy)
2. Patient who has a history of pallidotomy, thalamotomy, deep brain stimulation, or fetal tissue transplant
3. Patient who has dementia, active psychosis or hallucinations, or clinically significant depression
4. Patient who has a lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt), or has suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening
5. Patient who has a history of symptomatic orthostatic hypotension with a decrease of less than or equal to 20 mmHg in systolic blood pressure (SBP) or great than or equal to 10 mmHg in diastolic blood pressure when changing from supine to standing position after having been at supine position for at least 5 minutes within 28 days prior to the Screening Visit, or SBP less than 105 mmHg at study entry, or reports clinical signs of clinically significant orthostatic hypotension within 28 days prior to the Screening Visit.
6. Patient who is receiving therapy with a dopamine agonist either concurrently or has done so within 28 days prior to the Screening
7. Patient who is receiving therapy with 1 of the following drugs either concurrently or within 28 days prior to screening: MAO-B inhibitors, DA releasing agents, DA modulating agent, DA antagonists, neuroleptics, or other medications that may interact with DA function.
8. Patient who is currently receiving central nervous system active therapy (e.g., sedatives, hypnotics, antidepressants, anxiolytics), unless the dose has been stable for at least 28 days prior to Screening Visit and is likely to remain stable for the duration of the study. Patients should not take those medications within 8 hours prior to clinical visits
9. Patient who has a current diagnosis of epilepsy, has a history of seizures as an adult, has a history of stroke, or has had a transient ischemic attack within 1 year prior to Screening
10. Patient who has a history of known intolerance/hypersensitivity to non-dopaminegic antiemetics, such as domperidone, ondansetron, tropisetron, and glycopyrrolate
11. Patient who has any other clinically relevant hepatic, renal and cardiac dysfunction, or other medical condition or laboratory abnormality including abnormal plasma magnesium level, which would in the judgment of the investigator, interfere with the patient's ability to participate in the study
12. Patient who has a history of significant skin hypersensitivity to adhesive or other transdermal preparations or recent unresolved contact Dermatitis
13. Patient with C-reactive protein levels of 2x of upper limit of normal range
14. Female patient who is pregnant or is breastfeeding or is of childbearing potential without adequate contraception.
15. Patient with a positive finding in drug screening test or alcohol test

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-05; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
CMax of ROTIGOTINE | 38 Days
  PK parameters Cmax-ss

CONTACTS AND LOCATIONS:
Overall Officials: Simon Li, MD, Study Chair — Luye Pharma
Locations (3):
- United States (3):
  - CNS Network, Long Beach, California
  - MD Clinical, Hallandale, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No